CLINICAL TRIAL: NCT01028872
Title: Spherical Aberration and Contrast Sensitivity Function in Eyes Implanted With Spherical and Aspheric Intraocular Lenses: A Clinical Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Other Study IDs: 8547
Record Dates: First submitted 2009-12-08; First posted 2009-12-09 (Estimated); Last update posted 2009-12-09 (Estimated); Status verified 2006-09

CONDITIONS: Cataract
Keywords: higher-order aberrations, contrast sensitivity
MeSH Terms: conditions — Cataract | interventions — Lenses, Intraocular

ARMS (3):
- Sensar IOL (Sham Comparator)
  Interventions: Device: Intraocular lens
- Tecnis IOL (Active Comparator)
  Interventions: Device: Intraocular lens
- AcrySof IQ (Active Comparator)
  Interventions: Device: Intraocular lens

INTERVENTIONS:
Device: Intraocular lens
  Arms: Sensar IOL
Device: Intraocular lens
  Arms: Tecnis IOL
Device: Intraocular lens
  Arms: AcrySof IQ

SUMMARY:
Aspheric intraocular lenses can effectively reduce higher-order aberrations and improve contrast sensitivity function after cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* Senile cataract

Exclusion Criteria:

* Glaucoma, corneal opacity, retinal abnormality, previous history

Ages: 55 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Labbafinejad Medical Center, Tehran, Iran